CLINICAL TRIAL: NCT00133848
Title: A Randomised, Double-blind, Multicentre, Superiority Placebo-controlled, Phase III Study to Assess the Efficacy and Safety of Topical 1% SB-275833 Ointment Versus Placebo Ointment Applied Twice Daily for 5 Days in the Treatment of Adults and Paediatric Subjects With Impetigo.
Brief Title: Treatment Of Impetigo With Topical SB-275833 Ointment, 1% Versus Topical Placebo Ointment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: TOC103469
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Impetigo
Keywords: impetigo; topical antibacterial; topical antibiotic
MeSH Terms: conditions — Impetigo

INTERVENTIONS:
Drug: SB-275833 ointment, 1%
  Other Names: SB-275833 ointment; 1%

SUMMARY:
The goal of this study is to determine if topical SB-275833 ointment, 1% is more effective than a placebo ointment in the treatment of primary impetigo.

ELIGIBILITY:
Inclusion criteria:

* Must have primary impetigo with total lesion area being 100 square centimeters or less.
* Women who could bear children must have a negative urine pregnancy test and agree to either abstain from sexual intercourse or the use of specific effective contraceptive measures.

Exclusion Criteria:

* Any signs and symptoms of systemic infection.
* Any serious underlying disease that could be imminently life threatening.

Min Age: 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210
Dates: Start 2005-04; Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Clinical response of impetigo at end of therapy visit. Clinical response of success is defined as no further need for antibacterial treatment.

SECONDARY OUTCOMES:
Clinical response of impetigo at follow up visit. Impetigo lesion area at end of therapy and follow up visits.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (20):
- India (2):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Hyderabad
- GSK Investigational Site, Rome, Lazio, Italy
- Mexico (2):
  - GSK Investigational Site, Zapopan, Jalisco, Jalisco
  - GSK Investigational Site, Mexico City
- Netherlands (13):
  - GSK Investigational Site, Beek en Donk
  - GSK Investigational Site, Deurne
  - GSK Investigational Site, Ermelo
  - GSK Investigational Site, Gouda
  - GSK Investigational Site, Musselkanaal
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Nijverdal
  - GSK Investigational Site, Roelofarendsveen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Soerendonk
  - GSK Investigational Site, Woerden
  - GSK Investigational Site, Zieuwent
  - GSK Investigational Site, Zwijndrecht
- Peru (2):
  - GSK Investigational Site, Callao, Provincia Constitucional del Callao
  - GSK Investigational Site, Lima

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: TOC103469 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: TOC103469 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: TOC103469 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: TOC103469 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: TOC103469 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: TOC103469 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: TOC103469 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register